CLINICAL TRIAL: NCT07313306
Title: Feasibility of Symptom Management for Patients With Metastatic Breast Cancer to Increase Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC2513
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Metastatic Breast Cancer
Keywords: Get Real and Heel (GRH); physical activity; exercise; quality of life; social support
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — lime

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metastatic breast cancer (MBC) receive Get Real and Heel (GRH) (Experimental): Participants will receive Get Real and Heel (GRH) exercise program.
  Interventions: Behavioral: The Real and Heel (GRH)

INTERVENTIONS:
Behavioral: The Real and Heel (GRH) — The Get Real and Heel (GRH) program is a 16-week exercise intervention developed at the University of North Carolina at Chapel Hill (UNC).

SUMMARY:
This study will examine unmet exercise needs among patients with metastatic breast cancer (MBC) at UNC and assess whether participation in Get Real and Heel (GRH) can increase physical activity. The proposed research aims to improve multiple domains of well-being, quality of life, physical function, social support and reduce social isolation through a community based exercise intervention. By leveraging underutilized University of North Carolina Chapel Hill (UNC) resources, this work seeks to reduce barriers to accessibility, awareness, and appropriateness of exercise programming for this underserved population. Findings will help close the gap between patients' exercise needs, interest, and participation, with potential benefits for symptoms, functioning, and quality of life.

DETAILED DESCRIPTION:
Patients with MBC are living longer due to improved treatments, yet up to 92% experience functional decline and reduced quality of life. Exercise is a recommended, safe, and effective intervention for improving function, strength, fitness, and quality of life, but most patients do not meet guidelines. At UNC, a recent needs-assessment survey study of MBC patients (n=50) found that 52% were sedentary, although 72% believed increased exercise would improve treatment tolerance. GRH, established in 2006, offers 16 weeks of free, expert-led exercise including aerobic, strength, balance, and flexibility training tailored to participant needs. Despite its availability, only 4% of surveyed patients had been referred.

This study will evaluate the feasibility of implementing GRH for all MBC patients at UNC and assess its impact on quality of life, physical functioning, fatigue, and social isolation. Feasibility will be defined as attending ≥24 of 32 sessions. Patient-reported outcomes including Functional Assessment of Cancer Therapy- Breast (FACT-B), Patient-Reported Outcomes Measurement Information System (PROMIS) -Physical Function, the modified Medical Outcomes Social Support Survey, and PROMIS Social Isolation-will be collected electronically at baseline and at 16 weeks.

ELIGIBILITY:
In order to participate in this study a subject must meet all of the eligibility criteria outlined below.

Inclusion Criteria:

* Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
* Subjects are willing and able to comply with study procedures based on the judgement of the investigator or protocol designee.
* Age > 18 years at the time of consent.
* Diagnosis of metastatic breast cancer within two years of consent date
* Receives medical clearance from clinical team for moderate intensity exercise programming
* Indicates intent to receive ongoing cancer care at the enrolling institution
* English Speaking - program and measures are in English and not practicably translatable for a study this size.

Exclusion Criteria:

* Currently on hospice.
* Bed-bound status or other contraindication to exercise
* Participation in GRH since their diagnosis with MBC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of referral to Get Real and Heel | Up to 16 weeks
  The proportion of consented patients who are successfully referred to the Get Real and Heel program and complete at least 24 sessions (32 total available; 2 sessions per week) in person.

SECONDARY OUTCOMES:
Differences in quality of life - Functional Assessment of Cancer Therapy- Breast (The FACT-B) | 16 weeks
  Differences in quality of life will be measured from the baseline (start of Get Real and Heel program) and post-16-week follow-up Functional Assessment of Cancer Therapy- Breast (The FACT-B) scores. The FACT-B is a breast-cancer specific survey consisting of 37 questions regarding quality of life over the past 7 days. Total scores range 0-148. Higher scores indicate lower health-related quality of life.
Differences in quality of life - Patient Reported Outcomes Measurement Information System (PROMIS) -Physical Function | 16 weeks
  Differences in quality of life will be measured from the baseline (start of Get Real and Heel program) and post-16-week follow-up Patient Reported Outcomes Measurement Information System (PROMIS) -Physical Function 8c scores. The PROMIS Physical Function 8c asks about physical function over a 7-day period and is recommended to assess tolerance to drug therapy in the cancer population. The raw scores are then converted to a T-score, with higher scores indicating better function.
Differences in quality of life - Patient Reported Outcomes Measurement Information System (PROMIS) -Social Isolation | 16 weeks
  Differences in quality of life will be measured from the baseline (start of Get Real and Heel program) and post-16-week follow-up Patient Reported Outcomes Measurement Information System (PROMIS) -Social Isolation scores. The PROMIS Social Isolation survey asks about feelings of disconnection or exclusion from others where a T-score is utilized as a summary measure, with higher values indicating more social isolation
Differences in social support | 16 weeks
  Differences in social support will be measured from the baseline (start of GRH program) and post-16-week follow-up modified Medical Outcomes Social Support (mMOS-SS) scores. The mMOS-SS is an eight-item questionnaire asks about emotional and tangible social support that has been validated in the cancer population, including breast cancer, with a range of 8 to 40, with higher scores indicating more social support.

CONTACTS AND LOCATIONS:
Overall Officials: Sasha Knowlton, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comphrehensive Cancer Center at University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials